CLINICAL TRIAL: NCT01976234
Title: Infective Complication After Surgery and Transfusion of Allogenic RBC Fresh or Stored
Brief Title: Stored RBC Transfusion and Immonomodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Researcher, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 04121985
Record Dates: First submitted 2013-09-30; First posted 2013-11-05 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh group (Active Comparator): Fresh group will receive RBC stored for less than 14 days
  Interventions: Other: Fresh RBC
- Old group (Active Comparator): Old group will receive RBC stored for 14 days or more
  Interventions: Other: Old RBC

INTERVENTIONS:
Other: Fresh RBC — Patients will receive fresh blood only
  Arms: Fresh group
Other: Old RBC
  Other Names: Patients will receive blood stored for 14 days or more
  Arms: Old group

SUMMARY:
Transfusion of RBC is associated with post operative infections. Our hypothesis is that stored blood could be related with increased post operative infection risk. Surgical patients transfused during the operation or immediately after will be included in our study. Patients will receive fresh or old blood during the whole recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients transfused during or in 24h after surgical operation

Exclusion Criteria:

* Patients transfused during the 30 days before the operation
* Immunodepressed patients
* Infections during the 30 days before operations
* Emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of infections | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Savino Spadaro, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Sant'Anna Hospital, Ferrara, Ferrara, Italy

REFERENCES:
- [Result] Juffermans NP, Vlaar AP, Prins DJ, Goslings JC, Binnekade JM. The age of red blood cells is associated with bacterial infections in critically ill trauma patients. Blood Transfus. 2012 Jul;10(3):290-5. doi: 10.2450/2012.0068-11. Epub 2012 Feb 22. PMID 22395349